CLINICAL TRIAL: NCT01755689
Title: Immunogenicity and Safety Study of GSK Biologicals' Meningococcal Vaccine 134612 With or Without Co-administration of Cervarix and Boostrix in Female Adolescents and Young Adults at 9-25 Years of Age
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Meningococcal Vaccine With or Without Co-administration of Cervarix and Boostrix in Female Adolescents and Young Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113823; 2012-001876-13 (EudraCT Number)
Record Dates: First submitted 2012-12-13; First posted 2012-12-24 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2017-11

CONDITIONS: Infections, Meningococcal
Keywords: pertussis; Meningococcal meningitis; Meningococcal infections; HPV; Neisseria meningitidis; Vaccines, conjugate; tetanus; diphtheria; Meningococcal vaccines; Immunogenicity
MeSH Terms: conditions — Meningococcal Infections; Whooping Cough; Meningitis, Meningococcal; Tetanus; Diphtheria | interventions — human papillomavirus vaccine, L1 type 16, 18; Boostrix

ARMS (5):
- Nimenrix+Cervarix (1,2,7-Month) Group (Experimental): Subjects in this group received 1 dose of Nimenrix vaccine at Month 0 and 3 doses of Cervarix vaccine at Month 1, Month 2 and Month 7. Both vaccines were administered intramuscularly (IM) in the deltoid region of the arm.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Cervarix®
- Nimenrix+Cervarix (0,1,6-Month) Group (Experimental): Subjects in this group received 1 dose of Nimenrix vaccine at Month 0 and 3 doses of Cervarix vaccine at Month 0, Month 1 and Month 6. Both vaccines were administered intramuscularly (IM) in the deltoid region of the arm.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Cervarix®
- Cervarix Group (Experimental): Subjects in this group received 3 doses of Cervarix vaccine at Month 0, Month 1 and Month 6, administered intramuscularly (IM) in the deltoid region of the arm.
  Interventions: Biological: Cervarix®
- Nimenrix+Cervarix+Boostrix Group (Experimental): Subjects in this group received 1 dose each of Nimenrix and Boostrix vaccines at Month 0 and 3 doses of Cervarix vaccine at Month 0, Month 1 and Month 6. All vaccines were administered intramuscularly (IM) in the deltoid region of the arm.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Cervarix®; Biological: Boostrix®
- Boostrix+Cervarix Group (Experimental): Subjects in this group received 1 dose of Boostrix vaccine at Month 0 and 3 doses of Cervarix vaccine at Month 0, Month 1 and Month 6. Both vaccines were administered intramuscularly (IM) in the deltoid region of the arm.
  Interventions: Biological: Cervarix®; Biological: Boostrix®

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One dose administered intramuscularly (IM) in the deltoid of the right arm.
  Other Names: Nimenrix®
  Arms: Nimenrix+Cervarix (0,1,6-Month) Group; Nimenrix+Cervarix (1,2,7-Month) Group; Nimenrix+Cervarix+Boostrix Group
Biological: Cervarix® — Three doses administered intramuscularly (IM) in the deltoid of the left arm.
Biological: Boostrix® — One dose administered intramuscularly (IM) in the deltoid of the left arm.
  Arms: Boostrix+Cervarix Group; Nimenrix+Cervarix+Boostrix Group

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of GSK Biologicals' meningococcal vaccine GSK134612 (MenACWY-TT) co-administered with Cervarix as compared to MenACWY-TT and Cervarix administered alone and the co-administration of MenACWY-TT with Cervarix and Boostrix as compared to MenACWY-TT administered alone and Cervarix co-administered with Boostrix.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* A female between, and including, 9 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from parents/guardian of the subject and written informed assent obtained from the subject if the subject is less than legal age, or written informed consent obtained from the subject if the subject has achieved legal age. The legal age will be determined according to local regulations in each participating country.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will be ≥10 mg/day prednisone or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after each study dose of vaccine(s), with the exception of licensed inactivated influenza vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational product or a non-investigational vaccine/product.
* Previous vaccination with a meningococcal polysaccharide or conjugate vaccine within the last 10 years.
* History of meningococcal disease since birth.
* History of serious allergic reaction following any other DTP-containing vaccine or any component of the study vaccines.
* History of encephalopathy within seven days of administration of a previous pertussis antigen-containing vaccine that is not attributable to another identifiable cause.
* Persons who experienced an Arthus-type hypersensitivity reaction following a prior dose of tetanus-toxoid containing vaccine should not receive Boostrix unless at least 10 years have elapsed since the last dose of tetanus-toxoid containing vaccine.
* Previous vaccination with a tetanus-toxoid containing vaccine within the previous five years.
* Temperature of ≥ 40.5°C (105°F) within 48 hours of receipt of a previous dose of DTP vaccine (diphtheria-tetanus-whole cell pertussis [DTPw] and/or diphtheria-tetanus-acellular pertussis [DTaP]), not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of receipt of a previous dose of DTP vaccine.
* Seizures with or without fever within three days of a previous dose of DTP vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and history directed physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of any allergic disease/reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Progressive neurologic disorder, unstable neurologic conditions, uncontrolled epilepsy or progressive encephalopathy.
* History of any neurologic disorders or seizures. A history of ADHD or depression or a history of a single, simple febrile seizure does not exclude a subject.
* Major congenital defects or serious chronic illness.
* Previous history of Guillain-Barré Syndrome.
* Bleeding disorders, such as hemophilia or thrombocytopenia, or subjects on anti-coagulant therapy.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Previous administration of MPL or AS04 adjuvant.
* History of chronic alcohol consumption and/or drug abuse.
* Pregnant or lactating female.
* A subject planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Subjects must be at least three months post-pregnancy and not breastfeeding to enter the study.

Ages: 9 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1300 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2014-04-29 (Actual); Study Completion 2014-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Santo Domingo, Dominican Republic
- GSK Investigational Site, Tartu, Estonia
- GSK Investigational Site, Bangkok, Thailand

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Rivera L, Chanthavanich P, Poder A, Suryakiran PV, Jastorff A, Van der Wielen M. MenACWY-TT is immunogenic when co-administered with Tdap and AS04-HPV16/18 in girls and young women: Results from a phase III randomized trial. Vaccine. 2018 Jun 22;36(27):3967-3975. doi: 10.1016/j.vaccine.2018.05.051. Epub 2018 May 19. PMID 29789243

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Started | 259 | 259 | 261 | 260 | 261
Completed | 256 | 254 | 255 | 254 | 255
Not Completed | 3 | 5 | 6 | 6 | 6
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1 | 1
Not completed — Migrated/moved from study area | 0 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 2
Not completed — Pregnancy | 1 | 1 | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group | Total
Number analyzed (Participants) | 259 | 259 | 261 | 260 | 261 | 1300
Age, Continuous [Mean (Standard Deviation); unit: Participants] | 16.3 (4.6) | 16.6 (4.4) | 16.6 (4.6) | 16.6 (4.6) | 16.6 (4.5) | 16.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 259 | 261 | 260 | 261 | 1300
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage / African American | 0 | 0 | 0 | 1 | 0 | 1
  Geographic ancestry: Asian - South East Asian Heritage | 86 | 86 | 86 | 86 | 86 | 430
  Geographic ancestry: White - Caucasian / European Heritage | 87 | 86 | 87 | 87 | 88 | 435
  Geographic ancestry: Other | 86 | 87 | 88 | 86 | 87 | 434

OUTCOME MEASURES:

1. Primary Outcome: Anti-Meningitis Antibody Titers by Serum Bactericidal Assay Using Rabbit Complement (rSBA)
Description: The analysis was performed for the serogroups -MenA, -MenC -MenW-135 and -MenY. Antibody titers, tabulated as geometric mean titers (GMTs), were obtained by serum bactericidal assay using rabbit complement. This analysis was only performed on groups receiving Nimenrix vaccine.
Time Frame: At one month after vaccination with Nimenrix (Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination with Nimenrix.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Nimenrix+Cervarix+Boostrix Group
Number analyzed (Participants) | 256 | 255 | 257
Titers
  rSBA-MenA | 5517.1 [4791.4 to 6352.6] | 5523.5 [4913.2 to 6209.6] | 4649.6 [4022.8 to 5374.0]
  rSBA-MenC | 4277.3 [3604.3 to 5076.1] | 5091.0 [4338.6 to 5973.8] | 3598.6 [3004.2 to 4310.7]
  rSBA-MenW-135 | 14782.1 [12254.2 to 17831.5] | 18068.3 [15381.6 to 21224.4] | 11663.6 [9336.8 to 14570.2]
  rSBA-MenY | 11871.0 [10542.3 to 13367.2] | 12758.9 [11569.6 to 14070.5] | 11201.2 [9678.7 to 12963.1]
Statistical Analysis 1: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix+Boostrix Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix+Boostrix Group in terms of rSBA-MenA titers; Test type: Non-Inferiority — The non-inferiority criteria: the upper limit (UL) of the 2-sided standardised asymptotic 95% confidence interval (CI) for the ratio of rSBA GMTs had to be below the pre-defined limit of 2; ANCOVA; Adjusted GMT Ratio = 1.19, 95% CI 2-sided [0.99 to 1.43]
Statistical Analysis 2: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix (0,1,6-Month) Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix Group in terms of rSBA-MenA titers; Test type: Non-Inferiority — The non-inferiority criteria: the UL of the 2-sided standardised asymptotic 95% CI for the ratio of rSBA GMTs had to be below the pre-defined limit of 2; ANCOVA; Adjusted GMT Ratio = 1.01, 95% CI 2-sided [0.84 to 1.21]
Statistical Analysis 3: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix+Boostrix Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix+Boostrix Group in terms of rSBA-MenC titers; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; ANCOVA; Adjusted GMT Ratio = 1.19, 95% CI 2-sided [0.93 to 1.51]
Statistical Analysis 4: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix (0,1,6-Month) Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix Group in terms of rSBA-MenC titers; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; ANCOVA; Adjusted GMT Ratio = 0.83, 95% CI 2-sided [0.66 to 1.06]
Statistical Analysis 5: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix+Boostrix Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix+Boostrix Group in terms of rSBA-MenW-135 titers; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; ANCOVA; Adjusted GMT Ratio = 1.26, 95% CI 2-sided [0.97 to 1.64]
Statistical Analysis 6: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix (0,1,6-Month) Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix Group in terms of rSBA-MenW-135 titers; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; ANCOVA; Adjusted GMT Ratio = 0.82, 95% CI 2-sided [0.63 to 1.07]
Statistical Analysis 7: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix+Boostrix Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix+Boostrix Group in terms of rSBA-MenY titers; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; ANCOVA; Adjusted GMT Ratio = 1.05, 95% CI 2-sided [0.89 to 1.24]
Statistical Analysis 8: Comparison: Nimenrix+Cervarix (1,2,7-Month) Group vs Nimenrix+Cervarix (0,1,6-Month) Group; Adjusted GMT ratio of the Nimenrix Group versus Nimenrix+Cervarix Group in terms of rSBA-MenY titers; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; ANCOVA; Adjusted GMT Ratio = 0.95, 95% CI 2-sided [0.80 to 1.12]

2. Primary Outcome: Anti-HPV-16 and Anti-HPV-18 Concentrations
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as Enzyme-linked Immunosorbent Assay (ELISA) units per milliliter (EU/mL).
Time Frame: At one month after vaccination with Cervarix (Month 7)
Population: The analysis was performed on the ATP cohort for immunogenicity after Cervarix vaccination, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one HPV antigen component for the blood sample taken one month after the last Cervarix vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 248 | 249 | 244 | 247
EU/mL
  Anti-HPV-16 | 12124.9 [10564.5 to 13915.7] | 11672.1 [10173.5 to 13391.4] | 9563.8 [8262.0 to 11070.7] | 11470.7 [10018.5 to 13133.5]
  Anti-HPV-18 | 5234.1 [4573.9 to 5989.6] | 5655.0 [4978.5 to 6423.4] | 4306.2 [3748.3 to 4947.1] | 5110.0 [4487.0 to 5819.6]
Statistical Analysis 1: Comparison: Nimenrix+Cervarix (0,1,6-Month) Group vs Cervarix Group; Adjusted GMT ratio of the Cervarix Group versus Nimenrix+Cervarix (0,1,6-Month) Group in terms of HPV-16 titers; Test type: Non-Inferiority — For HPV-16, one month after the third dose of Cervarix, the UL of the two-sided standardized asymptotic 95% CI on the group GMT ratio had to be below the pre-defined limit of 2; ANCOVA; Adjusted GMT = 0.97, 95% CI 2-sided [0.81 to 1.15]
Statistical Analysis 2: Comparison: Nimenrix+Cervarix (0,1,6-Month) Group vs Cervarix Group; Adjusted GMT ratio of the Cervarix Group versus Nimenrix+Cervarix (0,1,6-Month) Group in terms of HPV-18 titers; Test type: Non-Inferiority — For HPV-18, one month after the third dose of Cervarix, the UL of the two-sided standardized asymptotic 95% CI on the group GMT ratio had to be below the pre-defined limit of 2; ANCOVA; Adjusted GMT = 1.09, 95% CI 2-sided [0.92 to 1.29]
Statistical Analysis 3: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; Adjusted GMT ratio of the Boostrix+Cervarix Group versus Nimenrix+Cervarix+Boostrix Group in terms of HPV-16 titers; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMT = 1.20, 95% CI 2-sided [1.01 to 1.43]
Statistical Analysis 4: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; Adjusted GMT ratio of the Boostrix+Cervarix Group versus Nimenrix+Cervarix+Boostrix Group in terms of HPV-18 titers; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; ANCOVA; Adjusted GMT = 1.19, 95% CI 2-sided [1.00 to 1.41]

3. Primary Outcome: Number of Subjects With Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Concentrations Equal to or Above (≥) 1.0 IU/mL
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as International Units per milliliter (IU/mL). This analysis was only performed on the groups receiving Boostrix vaccine.
Time Frame: At one month after Boostrix vaccination (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination with Boostrix.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 250 | 256
Participants
  Anti-D | 235 | 248
  Anti-T | 249 | 256
Statistical Analysis 1: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; The group difference of the Nimenrix+Cervarix+Boostrix Group and Boostrix+Cervarix Group in terms of Anti-D titers; Test type: Non-Inferiority — For anti-D the lower limit (LL) of the 2-sided standardised asymptotic 95% CI for the group difference (Nimenrix+Cervarix+Boostrix Group minus Boostrix +Cervarix Group) had to be greater than or equal to the pre-defined limit of -10%; Difference between groups = -2.88, 95% CI 2-sided [-6.90 to 0.81]
Statistical Analysis 2: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; The group difference of the Nimenrix+Cervarix+Boostrix Group and Boostrix+Cervarix Group in terms of Anti-T titers; Test type: Non-Inferiority — For anti-T the LL of the 2-sided standardised asymptotic 95% CI for the group difference (Nimenrix+Cervarix+Boostrix Group minus Boostrix +Cervarix Group) had to be greater than or equal to the pre-defined limit of -10%; Difference between groups = -0.40, 95% CI 2-sided [-2.23 to 1.08]

4. Primary Outcome: Anti-Pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: The antibody concentrations were tabulated as GMCs and expressed as IU/mL. GMCs were only analyzed in subjects receiving Boostrix vaccination.
Time Frame: At one month after Boostrix vaccination (Month 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 247 | 256
IU/mL
  Anti-PT: number analyzed (Participants) | 245 | 254
  Anti-PT | 52.9 [46.4 to 60.4] | 73.2 [65.0 to 82.5]
  Anti-FHA | 278.7 [249.5 to 311.2] | 472.4 [419.7 to 531.8]
  Anti-PRN: number analyzed (Participants) | 246 | 256
  Anti-PRN | 193.4 [159.0 to 235.1] | 318.6 [262.4 to 386.8]
Statistical Analysis 1: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; Adjusted GMT ratio of the Nimenrix+Cervarix+Boostrix Group versus Boostrix+ Cervarix Group in terms of anti-PRN titers; Test type: Non-Inferiority — For anti-PRN the UL of the 2-sided standardised asymptotic 95% CI for the adjusted group ratio of GMCs (Nimenrix+Cervarix+Boostrix Group/Boostrix+Cervarix Group) had to be less than or equal to the pre-defined limit of 1.5; ANCOVA; Adjusted GMT Ratio = 1.53, 95% CI 2-sided [1.25 to 1.87]
Statistical Analysis 2: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; Adjusted GMT ratio of the Nimenrix+Cervarix Group versus Boostrix+ Cervarix Group in terms of anti-FHA titers; Test type: Non-Inferiority — For anti-FHA the UL of the 2-sided standardised asymptotic 95% CI for the adjusted group ratio of GMCs (Nimenrix+Cervarix+Boostrix Group/Boostrix+Cervarix Group) had to be less than or equal to the pre-defined limit of 1.5; ANCOVA; Adjusted GMT Ratio = 1.65, 95% CI 2-sided [1.42 to 1.93]
Statistical Analysis 3: Comparison: Nimenrix+Cervarix+Boostrix Group vs Boostrix+Cervarix Group; Adjusted GMT ratio of the Nimenrix+Cervarix Group versus Boostrix+ Cervarix Group in terms of anti-PT titers; Test type: Non-Inferiority — For anti-PT the UL of the 2-sided standardised asymptotic 95% CI for the adjusted group ratio of GMCs (Nimenrix+Cervarix+Boostrix Group/Boostrix+Cervarix Group) had to be less than or equal to the pre-defined limit of 1.5; ANCOVA; Adjusted GMT Ratio = 1.39, 95% CI 2-sided [1.20 to 1.61]

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titres ≥ 1:8 and ≥ 1:128
Description: The number of subjects with rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY antibody titers ≥ 1:8 and ≥ 1:128 prior to and one month after vaccination with Nimenrix vaccine.
Time Frame: Prior to and one month after vaccination with Nimenrix (Months 0 and 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination with Nimenrix.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Nimenrix+Cervarix+Boostrix Group
Number analyzed (Participants) | 256 | 255 | 257
Participants
  rSBA-MenA ≥1:8, Month 0: number analyzed (Participants) | 256 | 255 | 255
  rSBA-MenA ≥1:8, Month 0 | 112 | 118 | 129
  rSBA-MenC ≥1:8, Month 0: number analyzed (Participants) | 255 | 255 | 255
  rSBA-MenC ≥1:8, Month 0 | 34 | 29 | 40
  rSBA-MenW-135 ≥1:8, Month 0: number analyzed (Participants) | 256 | 255 | 256
  rSBA-MenW-135 ≥1:8, Month 0 | 23 | 24 | 22
  rSBA-MenY ≥1:8, Month 0: number analyzed (Participants) | 255 | 255 | 256
  rSBA-MenY ≥1:8, Month 0 | 86 | 102 | 80
  rSBA-MenA ≥1:128, Month 0: number analyzed (Participants) | 256 | 255 | 255
  rSBA-MenA ≥1:128, Month 0 | 78 | 86 | 82
  rSBA-MenC ≥1:128, Month 0: number analyzed (Participants) | 255 | 255 | 255
  rSBA-MenC ≥1:128, Month 0 | 20 | 10 | 23
  rSBA-MenW-135 ≥1:128, Month 0: number analyzed (Participants) | 256 | 255 | 256
  rSBA-MenW-135 ≥1:128, Month 0 | 22 | 23 | 20
  rSBA-MenY ≥1:128, Month 0: number analyzed (Participants) | 255 | 255 | 256
  rSBA-MenY ≥1:128, Month 0 | 84 | 99 | 74
  rSBA-MenA ≥1:8, Month 1 | 255 | 255 | 255
  rSBA-MenC ≥1:8, Month 1 | 254 | 253 | 253
  rSBA-MenW-135 ≥1:8, Month 1 | 253 | 255 | 250
  rSBA-MenY ≥1:8, Month 1 | 256 | 255 | 255
  rSBA-MenA ≥1:128, Month 1 | 255 | 255 | 255
  rSBA-MenC ≥1:128, Month 1 | 254 | 252 | 252
  rSBA-MenW-135 ≥1:128, Month 1 | 253 | 255 | 250
  rSBA-MenY ≥1:128, Month 1 | 256 | 255 | 255

6. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Vaccine Response
Description: rSBA vaccine response for serogroups A, C, W-135 and Y was defined as:
  * For initially seronegative subjects (pre-vaccination titre below the cut-off of 1:8): number of subjects with rSBA antibody titres ≥ 1:32 one month after vaccination.
  * For initially seropositive subjects (pre-vaccination titre ≥ 1:8): number of subjects with rSBA antibody titres at least four times the pre-vaccination antibody titres, one month after vaccination.
Time Frame: At one month after Nimenrix vaccination (Month 1)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Nimenrix+Cervarix+Boostrix Group
Number analyzed (Participants) | 256 | 255 | 256
Participants
  rSBA-MenA: number analyzed (Participants) | 256 | 255 | 255
  rSBA-MenA | 240 | 235 | 230
  rSBA-MenC: number analyzed (Participants) | 255 | 255 | 255
  rSBA-MenC | 250 | 251 | 246
  rSBA-MenW-135 | 252 | 255 | 248
  rSBA-MenY: number analyzed (Participants) | 255 | 255 | 256
  rSBA-MenY | 245 | 253 | 251

7. Secondary Outcome: Number of Subjects With Anti-T Antibody Concentrations ≥ 0.1 IU/mL and ≥ 1.0 IU/mL
Description: The antibody concentrations were tabulated as GMCs and expressed as IU/mL, only for the Nimenrix+Cervarix (1,2,7-Month) Group.
Time Frame: Prior to and one month after vaccination with Nimenrix (Months 0 and 1)
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after Nimenrix vaccination,only for Nimenrix+Cervarix (1,2,7-Month) Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group
Number analyzed (Participants) | 255
Participants
  Anti-T ≥ 0.1 IU/mL, Month 0 | 236
  Anti-T ≥ 0.1 IU/mL, Month 1 | 255
  Anti-T ≥ 1 IU/mL, Month 0 | 151
  Anti-T ≥ 1 IU/mL, Month 1 | 253

8. Secondary Outcome: Anti-T Antibody Concentrations
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as international units per milliliter (IU/mL). This analysis was only performed for the Nimenrix+Cervarix (1,2,7-Month) Group.
Time Frame: Prior to and one month after vaccination with Nimenrix (Months 0 and 1)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group
Number analyzed (Participants) | 255
IU/mL
  Anti-T, Month 0 | 1.2 [1.0 to 1.4]
  Anti-T, Month 1 | 25.4 [22.8 to 28.3]

9. Secondary Outcome: Number of Subjects With Anti-HPV-16 Concentrations ≥ 19 EU/mL and Anti-HPV-18 Concentrations ≥ 18 EU/mL
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as ELISA units per milliliter (EU/mL).
Time Frame: Prior to the first dose and one month after the third dose of Cervarix [Month 0 and Month 7/Month 8 in Nimenrix+Cervarix (1,2,7-Month) Group]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix+Boostrix+Cervarix Group: Subjects in this group received 1 dose each of Nimenrix and Boostrix vaccines at Month 0 and 3 doses of Cervarix vaccine at Month 0, Month 1 and Month 6. All vaccines were administered intramuscularly (IM) in the deltoid region of the arm.
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Boostrix+Cervarix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 246 | 248 | 249 | 244 | 247
Participants
  Anti-HPV-16, Month 0 | 17 | 29 | 32 | 29 | 22
  Anti-HPV-16, Month 7/Month 8 | 245 | 248 | 249 | 244 | 247
  Anti-HPV-18, Month 0 | 11 | 12 | 17 | 14 | 14
  Anti-HPV-18, Month 7/Month 8 | 245 | 248 | 249 | 244 | 247

10. Secondary Outcome: Number of Subjects Seroconverted for Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Seroconversion rate is defined as the appearance of antibodies (i.e. titers greater than or equal to the cut-off value) in the serum of subjects who are seronegative before vaccination. The antibody concentrations were calculated as GMCs and expressed as EU/mL.
Time Frame: Prior to and one month after the third dose of Cervarix (Month 0 and Month 7/Month 8)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 235 | 236 | 232 | 230 | 233
Participants
  Anti-HPV-16, Month 0: number analyzed (Participants) | 229 | 219 | 217 | 215 | 225
  Anti-HPV-16, Month 0 | 0 | 0 | 0 | 0 | 0
  Anti-HPV-16, Month 7/Month 8: number analyzed (Participants) | 229 | 219 | 217 | 215 | 225
  Anti-HPV-16, Month 7/Month 8 | 228 | 219 | 217 | 215 | 225
  Anti-HPV-18, Month 0 | 0 | 0 | 0 | 0 | 0
  Anti-HPV-18, Month 7/Month 8 | 234 | 236 | 232 | 230 | 233

11. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Concentrations
Description: The antibody concentrations were calculated as GMCs and expressed as EU/mL, only for the Nimenrix+Cervarix (1,2,7-Month) Group.
Time Frame: Prior to and one month after the third dose of Cervarix (Months 0 and 8)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one HPV antigen component for the blood sample taken one month after the last Cervarix vaccination from the Nimenrix+Cervarix (1,2,7-Month) Group.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group
Number analyzed (Participants) | 246
EU/mL
  Anti-HPV-16, Month 0 | 10.9 [10.2 to 11.6]
  Anti-HPV-16, Month 8 | 11128.2 [9471.8 to 13074.4]
  Anti-HPV-18, Month 0 | 9.8 [9.3 to 10.4]
  Anti-HPV-18, Month 8 | 5357.0 [4550.2 to 6306.9]

12. Secondary Outcome: Booster Responses for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Booster responses to the PT, FHA and PRN antigens were defined as:
  * For initially seronegative subjects (antibody concentrations: < 2.046 IU/ml for anti-FHA, < 2.187 IU/ml for anti-PRN, < 2.693 IU/ml for anti-PT), antibody concentration ≥ 4*cut_off IU/ml at Month 1 post-vaccination;
  * For initially seropositive subjects (antibody concentrations: ≥ 2.046 IU/ml for anti-FHA, ≥ 2.187 IU/ml for anti-PRN, ≥ 2.693 IU/ml for anti-PT) with pre-vaccination antibody concentration < 4*cut_off IU/ml : antibody concentration at Month 1 ≥ 4 fold the pre-vaccination antibody concentration;
  * For initially seropositive subjects (antibody concentrations: ≥ 2.046 IU/ml for anti-FHA, ≥ 2.187 IU/ml for anti-PRN, ≥ 2.693 IU/ml for anti-PT) with pre-vaccination antibody concentration ≥ 4*cut_off IU/ml : antibody concentration at Month 1 ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: At one month after Boostrix vaccination (Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Boostrix+Cervarix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 247 | 256
Participants
  Anti-PT: number analyzed (Participants) | 245 | 254
  Anti-PT | 218 | 235
  Anti-FHA | 240 | 247
  Anti-PRN: number analyzed (Participants) | 246 | 256
  Anti-PRN | 231 | 248

13. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations ≥ 0.1 IU/mL
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as international units per milliliter (IU/mL).
Time Frame: Prior to and one month after Boostrix vaccination (Month 0 and Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 251 | 256
Participants
  Anti-D, Month 0: number analyzed (Participants) | 249 | 254
  Anti-D, Month 0 | 214 | 223
  Anti-D, Month 1: number analyzed (Participants) | 250 | 256
  Anti-D, Month 1 | 250 | 256
  Anti-T, Month 0 | 239 | 248
  Anti-T, Month 1: number analyzed (Participants) | 250 | 256
  Anti-T, Month 1 | 250 | 256

14. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: as for outcome 13
Time Frame: Prior to and one month after Boostrix vaccination (Months 0 and 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 251 | 256
IU/mL
  Anti-D, Month 0: number analyzed (Participants) | 249 | 254
  Anti-D, Month 0 | 0.5 [0.4 to 0.5] | 0.5 [0.4 to 0.6]
  Anti-D, Month 1: number analyzed (Participants) | 250 | 256
  Anti-D, Month 1 | 4.7 [4.2 to 5.2] | 6.6 [5.9 to 7.4]
  Anti-T, Month 0 | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.5]
  Anti-T, Month 1: number analyzed (Participants) | 250 | 256
  Anti-T, Month 1 | 25.9 [23.4 to 28.8] | 15.4 [14.1 to 16.9]

15. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations Equal to or Above the Cut-off Value
Description: The antibody concentrations were calculated as GMCs and expressed as IU/mL. Anti-PT assay cut-off=2.693 IU/mL, anti-FHA assay cut-off=2.046 IU/mL, anti-PRN assay cut-off=2.187 IU/mL.
Time Frame: Prior to and one month after Boostrix vaccination (Months 0 and 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 251 | 256
Participants
  Anti-PT, Month 0: number analyzed (Participants) | 249 | 254
  Anti-PT, Month 0 | 156 | 153
  Anti-PT, Month 1: number analyzed (Participants) | 245 | 254
  Anti-PT, Month 1 | 240 | 252
  Anti-FHA, Month 0 | 235 | 244
  Anti-FHA, Month 1: number analyzed (Participants) | 247 | 256
  Anti-FHA, Month 1 | 247 | 256
  Anti-PRN, Month 0: number analyzed (Participants) | 250 | 256
  Anti-PRN, Month 0 | 218 | 229
  Anti-PRN, Month 1: number analyzed (Participants) | 246 | 256
  Anti-PRN, Month 1 | 246 | 256

16. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, prevented normal every day activities. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Symptoms were presented by vaccination site. Some groups do not have results for "Dose 2" because solicited local symptoms were not collected for these subjects at the Dose 2 timepoint.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 259 | 257 | 259 | 260 | 261
Participants
  Any Pain (Nimenrix), Dose 1: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Any Pain (Nimenrix), Dose 1 | 152 | 140 |  | 156 |
  Grade 3 Pain (Nimenrix), Dose 1: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Grade 3 Pain (Nimenrix), Dose 1 | 4 | 3 |  | 7 |
  Any Pain (Boostrix), Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Any Pain (Boostrix), Dose 1 |  |  |  | 189 | 200
  Grade 3 Pain (Boostrix), Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Grade 3 Pain (Boostrix), Dose 1 |  |  |  | 21 | 15
  Any Pain (Cervarix), Dose 1: number analyzed (Participants) | 0 | 257 | 259 | 260 | 261
  Any Pain (Cervarix), Dose 1 |  | 213 | 205 | 217 | 221
  Grade 3 Pain (Cervarix), Dose 1: number analyzed (Participants) | 0 | 257 | 259 | 260 | 261
  Grade 3 Pain (Cervarix), Dose 1 |  | 8 | 11 | 23 | 18
  Any Redness (Nimenrix), Dose 1: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Any Redness (Nimenrix), Dose 1 | 57 | 42 |  | 54 |
  Grade 3 Redness (Nimenrix), Dose 1: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Grade 3 Redness (Nimenrix), Dose 1 | 4 | 2 |  | 0 |
  Any Redness (Boostrix), Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Any Redness (Boostrix), Dose 1 |  |  |  | 73 | 53
  Grade 3 Redness (Boostrix), Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Grade 3 Redness (Boostrix), Dose 1 |  |  |  | 2 | 4
  Any Redness (Cervarix), Dose 1: number analyzed (Participants) | 0 | 257 | 259 | 260 | 261
  Any Redness (Cervarix), Dose 1 |  | 56 | 54 | 62 | 48
  Grade 3 Redness (Cervarix), Dose 1: number analyzed (Participants) | 0 | 257 | 259 | 260 | 261
  Grade 3 Redness (Cervarix), Dose 1 |  | 0 | 0 | 1 | 0
  Any Swelling (Nimenrix), Dose 1: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Any Swelling (Nimenrix), Dose 1 | 40 | 34 |  | 58 |
  Grade 3 Swelling (Nimenrix), Dose 1: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Grade 3 Swelling (Nimenrix), Dose 1 | 1 | 1 |  | 5 |
  Any Swelling (Boostrix), Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Any Swelling (Boostrix), Dose 1 |  |  |  | 79 | 58
  Grade 3 Swelling (Boostrix), Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Grade 3 Swelling (Boostrix), Dose 1 |  |  |  | 5 | 7
  Any Swelling (Cervarix), Dose 1: number analyzed (Participants) | 0 | 257 | 259 | 260 | 261
  Any Swelling (Cervarix), Dose 1 |  | 42 | 37 | 64 | 55
  Grade 3 Swelling (Cervarix), Dose 1: number analyzed (Participants) | 0 | 257 | 259 | 260 | 261
  Grade 3 Swelling (Cervarix), Dose 1 |  | 1 | 1 | 1 | 5
  Any Pain (Nimenrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Grade 3 Pain (Nimenrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Any Pain (Boostrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Grade 3 Pain (Boostrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Any Pain (Cervarix), Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Pain (Cervarix), Dose 2 | 193 |  |  |  |
  Grade 3 Pain (Cervarix), Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Pain (Cervarix), Dose 2 | 15 |  |  |  |
  Any Redness (Nimenrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness (Nimenrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Any Redness (Boostrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness (Boostrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Any Redness (Cervarix), Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Redness (Cervarix), Dose 2 | 43 |  |  |  |
  Grade 3 Redness (Cervarix), Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Redness (Cervarix), Dose 2 | 0 |  |  |  |
  Any Swelling (Nimenrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Grade 3 Swelling (Nimenrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Any Swelling (Boostrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Grade 3 Swelling (Boostrix), Dose 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Any Swelling (Cervarix), Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Swelling (Cervarix), Dose 2 | 41 |  |  |  |
  Grade 3 Swelling (Cervarix), Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Swelling (Cervarix), Dose 2 | 1 |  |  |  |
  Any Pain (Nimenrix), Across doses: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Any Pain (Nimenrix), Across doses | 152 | 140 |  | 156 |
  Grade 3 Pain (Nimenrix), Across doses: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Grade 3 Pain (Nimenrix), Across doses | 4 | 3 |  | 7 |
  Any Pain (Boostrix), Across doses: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Any Pain (Boostrix), Across doses |  |  |  | 189 | 200
  Grade 3 Pain (Boostrix), Across doses: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Grade 3 Pain (Boostrix), Across doses |  |  |  | 21 | 15
  Any Pain (Cervarix), Across doses: number analyzed (Participants) | 258 | 257 | 259 | 260 | 261
  Any Pain (Cervarix), Across doses | 193 | 213 | 205 | 217 | 221
  Grade 3 Pain (Cervarix), Across doses: number analyzed (Participants) | 258 | 257 | 259 | 260 | 261
  Grade 3 Pain (Cervarix), Across doses | 15 | 8 | 11 | 23 | 18
  Any Redness (Nimenrix), Across doses: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Any Redness (Nimenrix), Across doses | 57 | 42 |  | 54 |
  Grade 3 Redness (Nimenrix), Across doses: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Grade 3 Redness (Nimenrix), Across doses | 4 | 2 |  | 0 |
  Any Redness (Boostrix), Across doses: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Any Redness (Boostrix), Across doses |  |  |  | 73 | 53
  Grade 3 Redness (Boostrix), Across doses: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Grade 3 Redness (Boostrix), Across doses |  |  |  | 2 | 4
  Any Redness (Cervarix), Across doses: number analyzed (Participants) | 258 | 257 | 259 | 260 | 261
  Any Redness (Cervarix), Across doses | 43 | 56 | 54 | 62 | 48
  Grade 3 Redness (Cervarix), Across doses: number analyzed (Participants) | 258 | 257 | 259 | 260 | 261
  Grade 3 Redness (Cervarix), Across doses | 0 | 0 | 0 | 1 | 0
  Any Swelling (Nimenrix), Across doses: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Any Swelling (Nimenrix), Across doses | 40 | 34 |  | 58 |
  Grade 3 Swelling (Nimenrix), Across doses: number analyzed (Participants) | 259 | 257 | 0 | 260 | 0
  Grade 3 Swelling (Nimenrix), Across doses | 1 | 1 |  | 5 |
  Any Swelling (Boostrix), Across doses: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Any Swelling (Boostrix), Across doses |  |  |  | 79 | 58
  Grade 3 Swelling (Boostrix), Across doses: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261
  Grade 3 Swelling (Boostrix), Across doses |  |  |  | 5 | 7
  Any Swelling (Cervarix), Across doses: number analyzed (Participants) | 258 | 257 | 259 | 260 | 261
  Any Swelling (Cervarix), Across doses | 41 | 42 | 37 | 64 | 55
  Grade 3 Swelling (Cervarix), Across doses: number analyzed (Participants) | 258 | 257 | 259 | 260 | 261
  Grade 3 Swelling (Cervarix), Across doses | 1 | 1 | 1 | 1 | 5

17. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, rash, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)] and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination. Some groups do not have results for "Dose 2" because solicited local symptoms were not collected for these subjects at the Dose 2 timepoint.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Boostrix+Cervarix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 259 | 257 | 259 | 260 | 261
Participants
  Any Arthralgia, Dose 1 | 23 | 18 | 13 | 36 | 23
  Grade 3 Arthralgia, Dose 1 | 0 | 1 | 1 | 1 | 4
  Related Arthralgia, Dose 1 | 23 | 18 | 13 | 34 | 23
  Any Fatigue, Dose 1 | 87 | 95 | 85 | 110 | 101
  Grade 3 Fatigue, Dose 1 | 2 | 4 | 2 | 8 | 5
  Related Fatigue, Dose 1 | 82 | 92 | 79 | 103 | 99
  Any Gastrointestinal, Dose 1 | 21 | 27 | 23 | 29 | 22
  Grade 3 Gastrointestinal, Dose 1 | 1 | 1 | 0 | 2 | 0
  Related Gastrointestinal, Dose 1 | 19 | 27 | 21 | 26 | 20
  Any Headache, Dose 1 | 82 | 94 | 78 | 99 | 95
  Grade 3 Headache, Dose 1 | 5 | 3 | 5 | 5 | 4
  Related Headache, Dose 1 | 81 | 89 | 73 | 92 | 85
  Any Myalgia, Dose 1 | 65 | 83 | 85 | 96 | 101
  Grade 3 Myalgia, Dose 1 | 0 | 4 | 6 | 9 | 9
  Related Myalgia, Dose 1 | 60 | 81 | 82 | 92 | 100
  Any Rash, Dose 1 | 4 | 8 | 8 | 6 | 6
  Grade 3 Rash, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Rash, Dose 1 | 1 | 6 | 7 | 6 | 4
  Any Fever, Dose 1 | 24 | 32 | 15 | 38 | 27
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 21 | 31 | 14 | 37 | 25
  Any Urticaria, Dose 1 | 0 | 4 | 4 | 5 | 5
  Grade 3 Urticaria, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Urticaria, Dose 1 | 0 | 3 | 4 | 5 | 3
  Any Arthralgia, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Arthralgia, Dose 2 | 18 |  |  |  |
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia, Dose 2 | 0 |  |  |  |
  Related Arthralgia, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Arthralgia, Dose 2 | 18 |  |  |  |
  Any Fatigue, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Fatigue, Dose 2 | 61 |  |  |  |
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Fatigue, Dose 2 | 2 |  |  |  |
  Related Fatigue, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Fatigue, Dose 2 | 58 |  |  |  |
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Gastrointestinal, Dose 2 | 10 |  |  |  |
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Gastrointestinal, Dose 2 | 1 |  |  |  |
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Gastrointestinal, Dose 2 | 8 |  |  |  |
  Any Headache, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Headache, Dose 2 | 58 |  |  |  |
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Headache, Dose 2 | 3 |  |  |  |
  Related Headache, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Headache, Dose 2 | 55 |  |  |  |
  Any Myalgia, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Myalgia, Dose 2 | 73 |  |  |  |
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Myalgia, Dose 2 | 4 |  |  |  |
  Related Myalgia, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Myalgia, Dose 2 | 72 |  |  |  |
  Any Rash, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Rash, Dose 2 | 3 |  |  |  |
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Rash, Dose 2 | 0 |  |  |  |
  Related Rash, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Rash, Dose 2 | 3 |  |  |  |
  Any Fever, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Fever, Dose 2 | 11 |  |  |  |
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Fever, Dose 2 | 0 |  |  |  |
  Related Fever, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Fever, Dose 2 | 10 |  |  |  |
  Any Urticaria, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Any Urticaria, Dose 2 | 2 |  |  |  |
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Grade 3 Urticaria, Dose 2 | 0 |  |  |  |
  Related Urticaria, Dose 2: number analyzed (Participants) | 258 | 0 | 0 | 0 | 0
  Related Urticaria, Dose 2 | 2 |  |  |  |
  Any Arthralgia, Across doses | 34 | 18 | 13 | 36 | 23
  Grade 3 Arthralgia, Across doses | 0 | 1 | 1 | 1 | 4
  Related Arthralgia, Across doses | 34 | 18 | 13 | 34 | 23
  Any Fatigue, Across doses | 105 | 95 | 85 | 110 | 101
  Grade 3 Fatigue, Across doses | 4 | 4 | 2 | 8 | 5
  Related Fatigue, Across doses | 98 | 92 | 79 | 103 | 99
  Any Gastrointestinal, Across doses | 26 | 27 | 23 | 29 | 22
  Grade 3 Gastrointestinal, Across doses | 2 | 1 | 0 | 2 | 0
  Related Gastrointestinal, Across doses | 23 | 27 | 21 | 26 | 20
  Any Headache, Across doses | 101 | 94 | 78 | 99 | 95
  Grade 3 Headache, Across doses | 8 | 3 | 5 | 5 | 4
  Related Headache, Across doses | 99 | 89 | 73 | 92 | 85
  Any Myalgia, Across doses | 95 | 83 | 85 | 96 | 101
  Grade 3 Myalgia, Across doses | 4 | 4 | 6 | 9 | 9
  Related Myalgia, Across doses | 91 | 81 | 82 | 92 | 100
  Any Rash, Across doses | 7 | 8 | 8 | 6 | 6
  Grade 3 Rash, Across doses | 0 | 0 | 0 | 0 | 0
  Related Rash, Across doses | 4 | 6 | 7 | 6 | 4
  Any Fever, Across doses | 34 | 32 | 15 | 38 | 27
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 0
  Related Fever, Across doses | 30 | 31 | 14 | 37 | 25
  Any Urticaria, Across doses | 2 | 4 | 4 | 5 | 5
  Grade 3 Urticaria, Across doses | 0 | 0 | 0 | 0 | 0
  Related Urticaria, Across doses | 2 | 3 | 4 | 5 | 3

18. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events AE(s)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 31-day (Days 0-30) period following vaccination with Nimenrix, Boostrix or the first dose of Cervarix
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 259 | 259 | 261 | 260 | 261
Participants | 37 | 35 | 35 | 42 | 39

19. Secondary Outcome: Number of Subjects With Serious Adverse Events SAE(s)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 8)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 259 | 259 | 261 | 260 | 261
Participants | 3 | 2 | 5 | 7 | 6

20. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (from Month 0 to Month 8)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 259 | 259 | 261 | 260 | 261
Participants | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With New Onset Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: During the entire study period (from Month 0 to Month 8)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
Number analyzed (Participants) | 259 | 259 | 261 | 260 | 261
Participants | 3 | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) period following each vaccination, Unsolicited AEs: during the 31-day (Days 0-30) period following each vaccination; SAEs: throughout the whole study period (from Month 0 up to Month 8).
Arm/Group | Nimenrix+Cervarix (1,2,7-Month) Group | Nimenrix+Cervarix (0,1,6-Month) Group | Cervarix Group | Nimenrix+Cervarix+Boostrix Group | Boostrix+Cervarix Group
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/259 | 0/261 | 0/260 | 1/261
Serious Adverse Events (participants affected / at risk) | 3/259 | 2/259 | 5/261 | 7/260 | 6/261
Other Adverse Events (participants affected / at risk) | 232/259 | 228/259 | 222/261 | 236/260 | 243/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix+Cervarix (1,2,7-Month) Group (N=259) | Nimenrix+Cervarix (0,1,6-Month) Group (N=259) | Cervarix Group (N=261) | Nimenrix+Cervarix+Boostrix Group (N=260) | Boostrix+Cervarix Group (N=261)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix+Cervarix (1,2,7-Month) Group (N=259) | Nimenrix+Cervarix (0,1,6-Month) Group (N=259) | Cervarix Group (N=261) | Nimenrix+Cervarix+Boostrix Group (N=260) | Boostrix+Cervarix Group (N=261)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (41) | 18 (18) | 13 (13) | 36 (36) | 23 (23)
Erythema (Skin and subcutaneous tissue disorders) | 78 (100) | 68 (68) | 54 (54) | 90 (90) | 64 (64)
Fatigue (General disorders) | 105 (148) | 95 (95) | 85 (85) | 110 (110) | 101 (101)
Gastrointestinal disorder (Gastrointestinal disorders) | 26 (31) | 27 (27) | 23 (23) | 29 (29) | 22 (22)
Headache (Nervous system disorders) | 103 (147) | 98 (99) | 78 (78) | 102 (107) | 98 (101)
Myalgia (Musculoskeletal and connective tissue disorders) | 95 (139) | 83 (83) | 85 (85) | 96 (96) | 101 (101)
Pain (General disorders) | 217 (345) | 220 (220) | 205 (205) | 228 (228) | 233 (233)
Pyrexia (General disorders) | 35 (36) | 33 (34) | 16 (16) | 39 (39) | 28 (28)
Swelling (General disorders) | 62 (81) | 54 (54) | 37 (37) | 98 (98) | 70 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.